CLINICAL TRIAL: NCT04451096
Title: Probiotics-prebiotic Fiber Therapy Improved Bowel Opening Frequency and Whole Gut Transit Time in Parkinson's Disease Patients With Constipation: A Randomised Controlled Study
Brief Title: Probiotics-prebiotic Fiber Therapy in Parkinson's Disease Patients With Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Dr Norlinah Mohamed Ibrahim, Professor, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FF-2018-387
Record Dates: First submitted 2020-06-19; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease; Constipation
Keywords: Parkinson's disease; Constipation; Probiotics; Prebiotic; Gut transit time; Motor outcome; NMSS; PDQ39; Randomised controlled trial
MeSH Terms: conditions — Parkinson Disease; Constipation | interventions — Probiotics; Prebiotics

STUDY DESIGN:
Intervention Model Description: placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic with prebiotic (Active Comparator): Drug: Probiotic sachet containing granulated multiple strains of Lactobacillus and Bifidobacterium, granulated fermented milk, lactose, fructo-oligosaccharide (FOS) with orange flavouring.
  Interventions: Dietary Supplement: Probiotics with prebiotic
- Placebo (Placebo Comparator): Drug : Placebo sachet of granulated milk, lactose and orange flavouring, without FOS or microbial cells which appeared similar to the probiotics
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics with prebiotic — Patients were instructed to consume one sachet twice daily mixed with a glass of water, before or after meals, for a duration of 8 weeks
  Other Names: Multistrain Probiotics with prebiotic
  Arms: Probiotic with prebiotic
Dietary Supplement: Placebo — Patients were instructed to consume one sachet twice daily mixed with a glass of water, before or after meals, for a duration of 8 weeks
  Other Names: Granulated milk products
  Arms: Placebo

SUMMARY:
A double blinded randomised placebo controlled trial to evaluate the efficacy of probiotics on constipation symptoms and whole gut transit time in patients with Parkinson's disease.PD patients with constipation were randomized to receive a multi-strain probiotic (Lactobacillus spp and Bifidobacterium spp at 30 X 109 CFU) with fructo-oligosaccaride (FOS) or placebo (fermented milk) twice daily for 8 weeks. Primary outcomes include changes in the presence of constipation symptoms using 9 items of Garrigues Questionnaire (GQ), which included an item on bowel opening frequency. Secondary and exploratory outcomes include whole gut transit time (WGTT), quality of life (PDQ39-SI), motor (MDS-UPDRS) and non-motor symptoms (NMSS).

DETAILED DESCRIPTION:
This was an eight-week double-blind, randomized placebo-controlled intervention study involving 55 idiopathic PD patients attending tertiary hospital. This study was conducted in accordance with good clinical practice as per Declaration of Helsinki and was approved by the institution's Research and Ethics Committee (FF-2018-387). Written informed consent was obtained from all particpants prior to enrollment.

Participants were included if they were aged 18 or older; were diagnosed with idiopathic PD in Hoehn and Yahr stages 1-4, and fulfilled the Rome III criteria for functional constipation which requires the presence of recurrent abdominal pain 3 days per month in the last 3 months, and symptom onset 6 months prior to diagnosis, with additional criteria below to be fulfilled, as adapted from Longstreth, et al12.

1. Must include two or more of the following:

   1. Straining during at least 25% of defecations
   2. Lumpy or hard stools in at least 25% of defecations
   3. Sensation of incomplete evacuation for at least 25% of defecations d. Sensation of anorectal obstruction/blockage for at least 25% of defecations

   e. Manual maneuvers to facilitate at least 25% of defecations (e.g, digital evacuation, support of the pelvic floor) f. Fewer than 3 defecations per week
2. Loose stools are rarely present without the use of laxatives
3. There are insufficient criteria for IBS

Participants were excluded if they had: a MMSE score of ≤ 21/30; a positive stool occult blood screening; a diagnosis of secondary parkinsonism; previous history of small and large bowel disease; prior history of gastrointestinal tract surgery; use of probiotics or antibiotics two weeks prior to baseline visit; been on medications such as antidepressants or anticholinergics; history of lactose intolerance; concomitant diagnosis of hypothyroidism and diabetes mellitus.

All participants were assessed at baseline and at 8 weeks following intervention for all outcome assessments. At baseline, additional data on demographics (age, sex, educational level), duration of PD, dopaminergic medication, Hoehn & Yahr Scoring during ON period, and the level of physical activity were recorded at baseline. A sedentary behaviour was defined as being physically active < 4 hours /week.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older; were diagnosed with idiopathic PD
* PD with Hoehn and Yahr stages 1-4,
* Fulfilled the Rome III criteria for functional constipation

Exclusion Criteria:

* MMSE score of ≤ 21/30
* Positive stool occult blood screening
* Diagnosis of secondary parkinsonism
* Previous history of small and large bowel disease
* History of gastrointestinal tract surgery
* Use of probiotics or antibiotics two weeks prior to baseline visit
* Been on medications such as antidepressants or anticholinergics
* History of lactose intolerance
* Concomitant diagnosis of hypothyroidism and diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-06 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
constipation symptoms | 8 weeks
  The presence of constipation symptoms at baseline and at 8 weeks evaluated by
  Garrigues Questionnaire (GQ).GQ is a 21-item self-reported screening questionnaire to detect the presence of constipation symptoms, using two different sets of four-point Likert scale responses.Although 12 items assess bowel habits, 9 items specifically assess constipation symptoms and were used in our evaluation: (i)Feeling of blockage in the anus;(ii) Need to press around anus/vagina to complete bowel movement; (iii) Spend >10 minutes to pass stool;(iv) Straining during bowel movement;(v) Feeling of hard stool;(vi) Feeling of incomplete emptying sensation; (vii)Bowel opening frequency;(viii) Frequency of oral laxative use;(ix) Frequency of enema use

SECONDARY OUTCOMES:
Whole Gut Transit Time (WGTT) in hours | 8 weeks
  WGTT was measured at baseline and at the end of 8 weeks, using red carmine capsule. The mean change in the WGTT (WGTT 8 weeks - WGTT baseline) was compared between the two groups.
Frequency of patients with constipation (Bowel motion < 3 per week) in percentage | 8 weeks
  Based on the stool diary, the percentage of patients who experienced less than 3 BM per week was calculated at baseline and at the end of study.
Movement Disorders Society- Unified Parkinson's Disease Rating Scale Part 11 | 8 weeks
  This measures the motor aspects of activity of daily living and consists of 13 items with scores between 0- 52. This instrument is given at baseline and 8 weeks. Lower score indicates low severity
Movement Disorders Society- Unified Parkinson's Disease Rating Scale Part 111 | 8 weeks
  This measures the seveirty of motor symptoms using 18 items (score 0-72). This instrument is given at baseline and 8 weeks. Lower score indicates low severity.
Non motor symptom score | 8 weeks
  Change in non-motor symptoms severity scores using the Non motor Symptom Scale (NMSS) which consists of 9 domains (cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucination, attention/memory, gastrointestinal tract, urinary, sexual function and miscellaneous.Score ranges from minimum of 3 to 360. Lower score indicates lower severity
Parkinsons Disease Quality of Life -39 Summary Index (PDQ39SI) | 8 weeks
  Change in PD9 39-SI which measure 8 domains of Quality of Life ( Lower score indicates better quality of life)
Weight in kilogram | 8 weeks
  Change in body weight measurement in Kg
Height in metres | Baseline
  Height will be measured in meters at baseline
Body Mass Index (kg/m2) | 8 weeks
  Weight and height will be combined to report BMI in kg/m^

CONTACTS AND LOCATIONS:
Overall Officials: Norlinah Mohamed Ibrahim, MBBChMRCP, Principal Investigator — National University of Malaysia
Locations (1):
- Hospital Canselor Tuanku Muhriz, UKM Medical Center, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Todd CL, Johnson EE, Stewart F, Wallace SA, Bryant A, Woodward S, Norton C. Conservative, physical and surgical interventions for managing faecal incontinence and constipation in adults with central neurological diseases. Cochrane Database Syst Rev. 2024 Oct 29;10(10):CD002115. doi: 10.1002/14651858.CD002115.pub6. PMID 39470206